CLINICAL TRIAL: NCT00554970
Title: A Randomized, Open Label, Active-Controlled, 4-Treatment, 2-Period, 2 Parallel Block Crossover Pharmacokinetic and Safety Study of 2 Doses of MAP0010 in Adult Asthmatics
Brief Title: A Study of 2 Doses of MAP0010 in Adult Asthmatics
Acronym: P202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAP0010-CL-P202
Record Dates: First submitted 2007-10-30; First posted 2007-11-07 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: Adult Asthmatics
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 then Treatment 2 (Other): Subjects received Treatment 1 in period 1 followed by a 7 day washout period and then Treatment 2 in period 2. Treatment 1 was a single dose of MAP0010 low dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 2 was a single dose of Pulmicort Respules® 0.25mg dose delivered by nebulization twice daily for 7 days as per protocol.
  Interventions: Drug: MAP0010 low dose; Drug: Budesonide inhalation suspension 0.25mg
- Treatment 2 then Treatment 1 (Other): Subjects received Treatment 2 in period 1 followed by a 7 day washout period and then Treatment 1 period 2. Treatment 1 was a single dose of MAP0010 low dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 2 was a single dose of Pulmicort Respules® 0.25mg dose delivered by nebulization twice daily for 7 days as per protocol.
  Interventions: Drug: MAP0010 low dose; Drug: Budesonide inhalation suspension 0.25mg
- Treatment 3 then Treatment 4 (Other): Subjects received Treatment 3 in period 1 followed by a 7 day washout period and then Treatment 4 period 2. Treatment 3 was a single dose of MAP0010 high dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 4 was a single dose of Pulmicort Respules® 0.5mg dose delivered by nebulization twice daily for 7 days as per protocol.
  Interventions: Drug: MAP0010 high dose; Drug: Budesonide inhalation suspension 0.5mg
- Treatment 4 then Treatment 3 (Other): Subjects received Treatment 4 in period 1 followed by a 7 day washout period and then Treatment 3 in period 2. Treatment 3 was a single dose of MAP0010 high dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 4 was a single dose of Pulmicort Respules® 0.5mg dose delivered by nebulization twice daily for 7 days as per protocol.
  Interventions: Drug: MAP0010 high dose; Drug: Budesonide inhalation suspension 0.5mg

INTERVENTIONS:
Drug: MAP0010 low dose — a single dose of MAP0010 low dose delivered by nebulization twice daily for 7 days as per protocol
  Arms: Treatment 1 then Treatment 2; Treatment 2 then Treatment 1
Drug: MAP0010 high dose — a single dose of MAP0010 high dose delivered by nebulization twice daily for 7 days as per protocol
  Arms: Treatment 3 then Treatment 4; Treatment 4 then Treatment 3
Drug: Budesonide inhalation suspension 0.25mg — a single dose of Pulmicort Respules® 0.25mg delivered by nebulization twice daily for 7 days as per protocol
  Other Names: Pulmicort Respules®
  Arms: Treatment 1 then Treatment 2; Treatment 2 then Treatment 1
Drug: Budesonide inhalation suspension 0.5mg — a single dose of Pulmicort Respules® 0.5mg dose delivered by nebulization twice daily for 7 days as per protocol
  Other Names: Pulmicort Respules®
  Arms: Treatment 3 then Treatment 4; Treatment 4 then Treatment 3

SUMMARY:
The purpose of this study is to examine the blood levels of two doses of MAP0010 (a corticosteroid) and two doses of an approved corticosteroid in adult asthma and safety with twice daily dosing over 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult asthmatics with mild to moderate persistent asthma.
* 18 to 45 (up to the 46th birthday) years of age.
* Documented diagnosis of asthma at least 3 months prior to Visit 1, per NIH/NHLBI, EPR-3 criteria.
* Able to withhold short-acting bronchodilators (e.g., albuterol or ipratropium bromide) for at least 4 hours prior to clinic visits.
* Baseline FEV1 greater than or equal to 50% of predicted normal.

Exclusion Criteria:

* Any other significant illness/abnormality
* A history of upper or lower respiratory tract infection within 2 weeks
* A history of acute or severe asthma attack requiring ICU admission or ventilatory support.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan
Locations (1):
- West Coast Clinical Trials Phase 2-4, LLC, Long Beach, California, United States

REFERENCES:
- See also: National Institutes of Health — http://www.nih.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 4-treatment, 2-period crossover study. Subjects were randomized to receive either Treatments 1 (MAP0010 low dose) and 2 (Pulmicort Respules® 0.25mg) or 3 (MAP0010 high dose) and 4 (Pulmicort Respules® 0.5mg). Subjects were randomized to the following sequences: Tx 1 then Tx 2, Tx 2 then Tx 1, Tx 3 then Tx 4, or Tx 4 then Tx 3
Groups:
- Treatment 2 Then Treatment 1: Subjects received Treatment 2 in period 1 followed by a 7 day washout period and then Treatment 1 in period 2. Treatment 1 was a single dose of MAP0010 low dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 2 was a single dose of Pulmicort Respules® 0.25mg dose delivered by nebulization twice daily for 7 days as per protocol.
- Treatment 3 Then Treatment 4: Subjects received Treatment 3 in period 1 followed by a 7 day washout period and then Treatment 4 in period 2. Treatment 3 was a single dose of MAP0010 high dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 4 was a single dose of Pulmicort Respules® 0.5mg dose delivered by nebulization twice daily for 7 days as per protocol.
Period: Period 1
Arm/Group | Treatment 1 Then Treatment 2 | Treatment 2 Then Treatment 1 | Treatment 3 Then Treatment 4 | Treatment 4 Then Treatment 3
Started | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8
Not Completed | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment 1 Then Treatment 2 | Treatment 2 Then Treatment 1 | Treatment 3 Then Treatment 4 | Treatment 4 Then Treatment 3
Started | 7 | 8 | 8 | 8
Completed | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment 2, Then Treatment 1: Subjects received Treatment 2 in period 1 followed by a 7 day washout period and then Treatment 1 in period 2. Treatment 1 was a single dose of MAP0010 low dose delivered by nebulization twice daily for 7 days as per protocol. Treatment 2 was a single dose of Pulmicort Respules® 0.25mg dose delivered by nebulization twice daily for 7 days as per protocol.
- Total: Total of all reporting groups
Arm/Group | Treatment 1 Then Treatment 2 | Treatment 2, Then Treatment 1 | Treatment 3 Then Treatment 4 | Treatment 4 Then Treatment 3 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (8.9) | 30.4 (7.2) | 30.0 (8.3) | 29.1 (6.9) | 29.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 7 | 19
  Male | 5 | 2 | 5 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Budesonide on Day 1 After Administration of MAP0010 Low Dose, MAP0010 High Dose, Pulmicort Respules® 0.25mg, and Pulmicort Respules® 0.5mg
Description: The maximum concentration (Cmax) is the highest concentration of a drug measured in the plasma. Plasma is the clear portion of the blood. The Cmax of Budesonide is reported in picograms per milliliter (pg/ml).
Time Frame: Day 1 hour 12
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Pulmicort Respules® 0.50 mg: a single dose of Pulmicort Respules® 0.5mg dose delivered by nebulization twice daily for 7 days as per protocol
- Pulmicort Respules® 0.25 mg: a single dose of Pulmicort Respules® 0.25mg dose delivered by nebulization twice daily for 7 days as per protocol
Arm/Group | MAP0010 High Dose | Pulmicort Respules® 0.50 mg | MAP0010 Low Dose | Pulmicort Respules® 0.25 mg
Number analyzed (Participants) | 16 | 16 | 16 | 15
pg/ml | 250 (161) | 365 (203) | 168 (130) | 197 (102)

2. Primary Outcome: Cmax of Budesonide on Day 8 After Administration of MAP0010 Low Dose, MAP0010 High Dose, Pulmicort Respules® 0.25mg, and Pulmicort Respules® 0.5mg
Description: as for outcome 1
Time Frame: Day 8 hour 12
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MAP0010 High Dose | Pulmicort Respules® 0.50 mg | MAP0010 Low Dose | Pulmicort Respules® 0.25 mg
Number analyzed (Participants) | 16 | 15 | 16 | 15
pg/ml | 528 (257) | 530 (334) | 366 (262) | 315 (206)

3. Primary Outcome: AUC(0-inf) of Budesonide on Day 1 After Administration of MAP0010 Low Dose, MAP0010 High Dose, Pulmicort Respules® 0.25mg, and Pulmicort Respules® 0.5mg
Description: The AUC(0-inf) is the area under the plot of plasma concentration of drug against time after drug administration. Budesonide AUC(0-inf) is reported in picograms times minutes per milliliter (pg*min/ml).
Time Frame: Day 1 hour 12
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | MAP0010 High Dose | Pulmicort Respules® 0.50 mg | MAP0010 Low Dose | Pulmicort Respules® 0.25 mg
Number analyzed (Participants) | 14 | 15 | 16 | 13
pg*min/ml | 19400 (7280) | 55900 (19800) | 10300 (4620) | 26900 (7420)

4. Primary Outcome: AUC(0-inf) of Budesonide on Day 8 After Administration of MAP0010 Low Dose, MAP0010 High Dose, Pulmicort Respules® 0.25mg, and Pulmicort Respules® 0.5mg
Description: as for outcome 3
Time Frame: Day 8 hour 12
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | MAP0010 High Dose | Pulmicort Respules® 0.50 mg | MAP0010 Low Dose | Pulmicort Respules® 0.25 mg
Number analyzed (Participants) | 14 | 14 | 16 | 14
pg*min/ml | 58700 (25700) | 90100 (38200) | 35500 (15000) | 45200 (19500)

5. Primary Outcome: Half-life (t1/2) of Budesonide on Day 1 After Administration of MAP0010 Low Dose, MAP0010 High Dose, Pulmicort Respules® 0.25mg, and Pulmicort Respules® 0.5mg
Description: Half-life (t1/2) is the time for the drug to decrease to half of its maximum concentration. Budesonide t1/2 is reported in minutes.
Time Frame: Day 1 hour 12
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | MAP0010 High Dose | Pulmicort Respules® 0.50 mg | MAP0010 Low Dose | Pulmicort Respules® 0.25 mg
Number analyzed (Participants) | 14 | 15 | 16 | 13
min | 168 (95.7) | 207 (110) | 112 (49.0) | 179 (75.8)

6. Primary Outcome: Half-life (t1/2) of Budesonide on Day 8 After Administration of MAP0010 Low Dose, MAP0010 High Dose, Pulmicort Respules® 0.25mg, and Pulmicort Respules® 0.5mg
Description: as for outcome 5
Time Frame: Day 8 hour 12
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | MAP0010 High Dose | Pulmicort Respules® 0.50 mg | MAP0010 Low Dose | Pulmicort Respules® 0.25 mg
Number analyzed (Participants) | 14 | 14 | 16 | 14
min | 193 (67.2) | 192 (66.3) | 248 (192) | 230 (130)

ADVERSE EVENTS:
Description: Adverse events are presented by treatment arm, not by individual treatment (intervention) received.
Arm/Group | Treatment 1 Then Treatment 2 | Treatment 2, Then Treatment 1 | Treatment 3 Then Treatment 4 | Treatment 4 Then Treatment 3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 2/8 | 3/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 Then Treatment 2 (N=8) | Treatment 2, Then Treatment 1 (N=8) | Treatment 3 Then Treatment 4 (N=8) | Treatment 4 Then Treatment 3 (N=8)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal polyps (Nervous system disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.